CLINICAL TRIAL: NCT04807777
Title: A Multi-Center Phase II Study of Ruxolitinib in Solid Organ Transplant Recipients With Advanced Cutaneous Squamous Cell Carcinoma
Brief Title: Study of Ruxolitinib in Solid Organ Transplant Recipients With Advanced Cutaneous Squamous Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Departure of the original investigator
Sponsor: Columbia University (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Principal Investigator, Alexander Z. Wei, MD, Assistant Professor of Medicine at the Columbia University Medical Center, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAT5353
Record Dates: First submitted 2021-01-08; First posted 2021-03-19 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Advanced Cutaneous Squamous Cell Carcinoma
Keywords: Ruxolitinib; Solid Organ Transplant
MeSH Terms: interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ruxolitinib (Experimental): In a safety lead-in of 6 patients, subjects will receive 15mg of ruxolitinib twice daily (BID). After 4 weeks, if dose-limiting toxicities (DLT) are observed in 1 or fewer patients, the study will enter stage 1 of the Simon two-stage design where all subsequent patients will receive a starting dose of ruxolitinib 15mg BID.
  Subjects will have regularly scheduled study visits at the clinical site on Day 1 and Day 15 (± 3 days) of the first 2 cycles, then on Day 1 (± 3 days) of every subsequent cycle (starting cycle 3), where safety assessments, including laboratory assessments, vital signs, and physical examinations will be performed.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib will be administered orally twice daily during the entirety of each 28-day cycle.
  Other Names: JAKAVI

SUMMARY:
In this open-label, multicenter, Phase II study, the investigators propose to evaluate the efficacy of ruxolitinib, an orally administered inhibitor of JAK1/2, in solid organ transplant recipients with advanced cSCC. In a safety lead-in of 6 patients, subjects will receive ruxolitinib 15mg twice daily (BID). After 4 weeks, if dose-limiting toxicities (DLT) are observed in 1 or fewer patients, the study will enter stage 1 of the Simon two-stage design where all subsequent patients will receive a starting dose of ruxolitinib 15mg BID. If more than 1 DLTs are observed, another cohort of 6 patients will be treated at a dose of 10mg BID. If less than 2 DLTs are observed at the new dose of 10mg, then the study will proceed to stage I using this dose; otherwise the study will stop.

DETAILED DESCRIPTION:
Approximately 5.4 million individuals in the United States are diagnosed with non-melanoma skin cancers (NMSC) annually, with the incidence increasing over time. Twenty-five percent are cutaneous squamous cell carcinomas (cSCC), which affect up to 1,350,000 individuals and result in up to 12,000 deaths annually in the US alone. Immunosuppressed patients are particularly vulnerable to the development of highly aggressive or catastrophic cSCC. Patients receiving immunosuppressive therapy, such as solid organ transplant recipients (SOTRs), and HIV/AIDS patients have an estimated 60 to 250-fold increased risk of cSCC development. In renal SOTRs, cSCC represents over 70% of all malignancies that develop, with an incidence up to 200 times that of the general population. Post-transplant cSCC occurs at a younger age and is more aggressive than in non-transplant cohorts, with 30% of cSCC recurring within 1 year and up to 8% of disease associated with metastasis. The median survival from diagnosis of metastasis is 3 years.5 Cemiplimab, an anti-PD1 antibody, recently became the first agent to achieve regulatory approval for the treatment of advanced cSCC; however, due to the risk of graft rejection, the role of immunological checkpoint blockade in the SOTR population is extremely limited. Thus, although surgical excision is effective for sporadic cSCC, there remains a large unmet medical need for novel strategies for treatment and/or prevention of multiply recurrent, locally advanced, and metastatic cSCC, particularly in immunosuppressed patients.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed diagnosis of metastatic advanced cutaneous squamous cell carcinoma.
* History of solid-organ transplant requiring immunosuppression
* Age ≥ 18 yrs
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Karnofsky Performance Status Scale (KPS) ≥60%, Eastern Cooperative Oncology Group (ECOG) ≤2
* No prior Janus kinase (JAK) Inhibitor therapy
* Adequate organ function
* All clinically significant toxicities from prior systemic therapy must be ≤ Grade 1 (with the exception of alopecia, and peripheral neuropathy, which may be ≤ grade 2).
* Subjects must agree to undergo tumor biopsies until biopsies have been obtained from 10 subjects (i.e., biopsies are required in at least the first 10 enrolled subjects, or until a goal of 10 study biopsies are obtained). Subjects in whom a biopsy is technically not feasible or in whom would result in unacceptable risk in the opinion of the investigator, may be exempted from the biopsy requirement with discussion with the principal investigator.
* Negative pregnancy test for women of child bearing potential
* Ability to take oral medications
* Adequate marrow function:

  * Absolute neutrophil count (ANC) ≥1000 /mm3
  * Platelet count ≥50,000/mm3
  * Hemoglobin ≥8.0g/dL (not requiring transfusion in the past 2 weeks)

Exclusion Criteria:

* At least 21 days must have elapsed since the last dose of systemic chemotherapy or immunotherapy and the first dose of study drug.
* At least 14 days must have elapsed since the last dose of radiation therapy and the first dose of study drug.
* Patients who have previously been treated with a JAK inhibitor.
* Patients who are receiving any other investigational agents concurrently.
* Patients who have had recent major surgery within a minimum 4 weeks prior to starting study treatment, with the exception of surgical placement for vascular access.
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to ruxolitinib.
* Patients with symptomatic or growing brain metastases. Patients with brain metastases that have been treated and have remained stable for at least one month prior to initiation of study therapy are eligible.
* Concurrent use of strong CYP3A4 or CYP3A4 substrate drugs with a narrow therapeutic range within 14 days or 5 drug half-lives, whichever is longer, before start of study drug. A list of strong CYP3A4 and 2C8 inhibitors and inducers can be found in Appendix A.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with ruxolitinib. In addition, these patients are at increased risk of lethal infections when treated with marrow- suppressive therapy.
* Subjects with known active hepatitis B or C, or chronic hepatitis B or C requiring treatment with antiviral therapy.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients being actively treated for a second malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Wei, MD, Principal Investigator — Associate Professor of Medicine at the Columbia University Medical Center
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

REFERENCES:
- See also: Columbia University Medical Center — https://www.cuimc.columbia.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Ruxolitinib: In a safety lead-in of 6 patients, subjects will receive 15mg of ruxolitinib twice daily (BID). After 4 weeks, if dose-limiting toxicities (DLT) are observed in 1 or fewer patients, the study will enter stage 1 of the Simon two-stage design where all subsequent patients will receive a starting dose of ruxolitinib 15mg BID.
  Subjects will have regularly scheduled study visits at the clinical site on Day 1 and Day 15 (± 3 days) of the first 2 cycles, then on Day 1 (± 3 days) of every subsequent cycle (starting cycle 3), where safety assessments, including laboratory assessments, vital signs, and physical examinations will be performed.
  Ruxolitinib: Ruxolitinib will be administered orally twice daily during the entirety of each 28-day cycle.
Period: Safety Lead-in: Ruxolitinib 15mg
Arm/Group | Ruxolitinib
Started | 3
Completed | 3
Not Completed | 0
Period: Stage 1
Arm/Group | Ruxolitinib
Started | 0 (The protocol specifies that 6 participants are to complete the safety lead in phase prior to moving onto stage 1 of the study. As the safety lead-in stage was not completed (only 3 participants were enrolled), stage 1 was not initiated.)
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: The primary endpoint is the overall response rate as defined as the best response, confirmed at ≥4 weeks using RECIST v1.1 criteria. Responses defined as: Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions). Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: within the first 24 weeks of the start of study therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 3
Participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 1
  Progressive Disease | 2

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival (PFS) (time alive without advanced cutaneous squamous cell carcinoma (cSCC) probabilities will be estimated
Time Frame: Up to 14 months
Measure: Mean (Full Range); unit: Days
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 3
Days | 46.67 [28 to 56]

3. Secondary Outcome: Overall Survival (OS)
Description: The length of time from the start of treatment that subjects with the disease are still alive.
Time Frame: Up to17 months
Measure: Mean (Full Range); unit: Days
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 3
Days | 290.67 [160 to 506]

ADVERSE EVENTS:
Time Frame: Up to 17 months
Description: Systematic collection of adverse events on Day 1 and Day 15 (± 3 days) of the first cycle, then on Day 1 (± 3 days) of every subsequent cycle (starting cycle 2).
Arm/Group | Ruxolitinib
All-Cause Mortality (participants affected / at risk) | 3/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib (N=3)
Anemia (Blood and lymphatic system disorders) | 1
Lung Infection (Infections and infestations) | 1
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Fatigue (General disorders) | 1
Flu like symptoms (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither the complete nor any part of the results of the study carried out under this protocol, nor any of the information provided by the sponsor for the purposes of performing the study, will be published or passed on to any third party without the consent of the study sponsor-investigator.

Any investigator involved with this study is obligated to provide the sponsor-investigator with complete test results and all data derived from the study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT04807777/Prot_SAP_000.pdf